CLINICAL TRIAL: NCT07009769
Title: Retrospective Clinical Study for Developing an AI-Driven Precision Diagnostic System for Lung Cancer Based on Liquid Biopsy
Brief Title: AI-Driven Precision Diagnostic System for Lung Cancer Based on Liquid Biopsy
Status: Completed | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hyun Koo Kim, Professor, Korea University Guro Hospital
Other Study IDs: 2024GR0131
Record Dates: First submitted 2025-05-29; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to develop an AI-powered precision medicine system based on liquid biopsy that can comprehensively provide lung cancer patients with information on disease stage, histologic subtype, and presence of genetic mutations.

ELIGIBILITY:
Inclusion Criteria (Patients)

* Republic of Korea nationality
* Age ≥ 30 years
* Lung cancer based on radiologic and/or histopathologic examination
* No prior diagnosis of any other cancer and no history of anticancer treatment before the date of blood sample collection

Exclusion Criteria (Patients)

* History of other cancers before blood collection
* Prior cancer treatment before blood collection
* Incomplete clinical data
* No consent for sample use

Inclusion Criteria (Healthy Controls):

* Republic of Korea nationality
* No history of any cancer
* Age ≥ 30 years

Exclusion Criteria (Healthy Controls):

* History of any malignancy
* Incomplete clinical information or no consent for sample use

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult lung cancer patients (≥18 years old) and healthy controls, all South Korean nationals, with plasma collected before any cancer treatment.
Sampling Method: Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the AI-based classification model using SERS signals from plasma-derived exosomes | Retrospective, based on pre-collected samples through study completion, an average of 1 year
  To evaluate the diagnostic performance (sensitivity, specificity, and overall accuracy) of a machine learning model trained on SERS spectral data of plasma-derived exosomes in distinguishing lung cancer patients from healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Guro-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
IPD will not be shared because the data contain sensitive clinical information, and current institutional and ethical guidelines prohibit public sharing of identifiable or potentially re-identifiable participant-level data.